CLINICAL TRIAL: NCT03123900
Title: Neuroplasticity in Adulthood: Physical Exercise and Cognitive Training; Integrative Omics Study on the Neurobiological Effects of Physical Activity and Cognitive Stimulation
Brief Title: Effects of Physical and Cognitive Training in Neuroplasticity, Health and Cognition. Movement Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Barcelona (Other)
Collaborators: Ministerio de Economía y Competitividad, Spain (Other Government); Fundacio d'Investigacio en Atencio Primaria Jordi Gol i Gurina (Other); Universitat Politècnica de Catalunya (Other); Institut Guttmann (Other); Germans Trias i Pujol Hospital (Other); University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Maria Mataro Serrat, PhD. Associate professor, University of Barcelona
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: PSI2013-47724P; PSI2016-77475R (Other Grant/Funding Number: Ministry of Economy and Competitiveness)
Record Dates: First submitted 2017-03-06; First posted 2017-04-21 (Actual); Last update posted 2018-10-23 (Actual); Status verified 2018-10

CONDITIONS: Aging; Cognitive Function 1, Social
MeSH Terms: interventions — Exercise; Cognitive Training

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Physical exercise (n= 40) (Experimental): Walking program up to 45 minutes, 5 times a week for 3 months.
  Interventions: Behavioral: Physical exercise
- Cognitive training (n=40) (Experimental): Computerized cognitive training up to 45 minutes, 5 times a week for 3 months.
  Interventions: Behavioral: Cognitive training
- Combined training (n=40) (Experimental): Exercise and cognitive training up to 90 minutes, 5 times a week for 3 months.
  Interventions: Behavioral: Combined training
- Control group (n=20) (No Intervention): Waiting list group.They receive no intervention during this waiting period. At the end of this period our training programs are available to them.

INTERVENTIONS:
Behavioral: Physical exercise — The structured physical activity plan consists of a walking program with an initial progressive phase (first week: 30 minutes/session and second week: 45 minutes/session, with a Borg scale of perceived exertion between 9 and 10) and an improvement and maintenance phase (10 weeks, 45 minutes/session with a Borg scale of perceived exertion between 11 and 14).
  Arms: Physical exercise (n= 40)
Behavioral: Cognitive training — We use a computerized cognitive training tele-medicine tool, designed by the Guttmann Institute: Guttmann Neuro Personal Trainer (PREVIRNET). Sessions will consist in activities of attention, memory and executive functions, also put in place progressively and parallel to the physical activity.
  Arms: Cognitive training (n=40)
Behavioral: Combined training — Subjects included in this group receive both types of intervention.
  Arms: Combined training (n=40)

SUMMARY:
The MoveMent project applies non-pharmacological strategies - physical exercise and cognitive training - that have been shown to be effective in promoting active and healthy aging. The objective is to study the molecular and neural mechanisms of these strategies to stimulate brain plasticity and improve brain health and cognitive functioning.

DETAILED DESCRIPTION:
It is a randomized controlled study with three intervention groups - physical, cognitive and combined - and a control group. The intervention is carried out over 3 months, with a frequency of 5 weekly sessions of 45 minutes each. Cognitive training is applied through a computerized program, physical training consists of a walking aerobic program, and combined training arises from the addition of the two previous ones.

140 participants will undergo an exhaustive pre- and post-intervention evaluation that includes neuropsychological, neuroimaging, genetic and biochemical analysis before and after the intervention as well as physical and health status assessment.

The present project aims to examine the independent and combined effects of exercise and cognitive stimulation in functional and structural brain plasticity, cognitive performance, emotional state and quality of life, and will determine the demographic and clinical factors that can modulate neuroplasticity. It will allow us to study the neurophysiological mechanisms by which the different types of intervention have an effect on the structure and functioning of the brain and cognition within an omics framework.

ELIGIBILITY:
Inclusion Criteria:

* Age between 50 and 70
* Underactive or sedentary (<2 hours a week of physical activity).
* Adequate visual, auditory and fine motor skills.
* Able to speak and understand Catalan or Spanish language.
* Accept to take part in the study and sign the informed consent according to the Declaration of Helsinki.

Exclusion Criteria:

* Mini mental State examination < 24 and Montreal Cognitive Assessment- Short (MoCA -S) < 6.
* Diagnosis of mild cognitive impairment, dementia or other serious neurological, psychiatric, or systemic illness.
* Presence of another illness that render them unable to engage in physical activity (signs or symptoms of chronic heart disease, chronic obstructive pulmonary disease, orthopedic problems).
* History of drug abuse or alcoholism.
* Psychotropic consumption
* Contraindication to magnetic resonance imaging

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2015-11-26 (Actual); Primary Completion 2018-04-08 (Actual); Study Completion 2018-04-08 (Actual)

PRIMARY OUTCOMES:
Changes in functional and structural brain plasticity assessed with Magnetic Resonance Imaging | Baseline and 3 months
  Resting state connectivity, structural connectivity, white matter integrity, tractography, volume of white and grey matter structures.

SECONDARY OUTCOMES:
Changes in cognitive function | Baseline and 3 months
  Tests of executive function, attention, memory, language, visuospatial abilities and speed
Changes in emotional and functional status: Cognitive decline | Baseline and 3 months
  Short Form of the Informant Questionnaire on Cognitive Decline in the Elderly (Short IQCODE)
Changes in emotional and functional status: Depression | Baseline and 3 months
  Geriatric Depression Scale (GDS)
Changes in emotional and functional status: Mood | Baseline and 3 months
  Adapted Visual Analog Mood Scale (VAMS)
Changes in emotional and functional status: Clinical outcome | Baseline and 3 months
  Spanish version of the Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM)
Changes in health, fitness and physical activity: Cardiovascular risk factors | Baseline and 3 months
  Cardiovascular risk factors
Changes in health, fitness and physical activity: Sleep | Baseline and 3 months
  Pittsburgh Sleep quality Index
Changes in health, fitness and physical activity: Physical activity questionnaire | Baseline and 3 months
  Spanish version of the reduced Minnesota leisure time physical and activity questionnaire (VREM)
Changes in health, fitness and physical activity: Fitness | Baseline and 3 months
  One-mile Rockport walk test
Changes in health, fitness and physical activity: Physical activity monitoring | Baseline and 3 months
  Polar Loop activity monitoring device.
Changes in metabolites and gene expression patterns | Baseline and 3 months
  Metabolomic and transcriptomic analyses

OTHER OUTCOMES:
Changes in global cognitive function | Baseline and 3 months
  Mini mental state examination

CONTACTS AND LOCATIONS:
Overall Officials: Maria Mataro Serrat, Ph.D., Principal Investigator — University of Barcelona
Locations (1):
- Centre Atenció Primària el Maresme, Mataró, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Roig-Coll F, Castells-Sanchez A, Lamonja-Vicente N, Toran-Monserrat P, Pera G, Garcia-Molina A, Tormos JM, Montero-Alia P, Alzamora MT, Dacosta-Aguayo R, Soriano-Raya JJ, Caceres C, Erickson KI, Mataro M. Effects of Aerobic Exercise, Cognitive and Combined Training on Cognition in Physically Inactive Healthy Late-Middle-Aged Adults: The Projecte Moviment Randomized Controlled Trial. Front Aging Neurosci. 2020 Oct 29;12:590168. doi: 10.3389/fnagi.2020.590168. eCollection 2020. PMID 33192485
- [Derived] Castells-Sanchez A, Roig-Coll F, Lamonja-Vicente N, Altes-Magret M, Toran-Monserrat P, Via M, Garcia-Molina A, Tormos JM, Heras A, Alzamora MT, Fores R, Pera G, Dacosta-Aguayo R, Soriano-Raya JJ, Caceres C, Montero-Alia P, Montero-Alia JJ, Jimenez-Gonzalez MM, Hernandez-Perez M, Perera A, Grove GA, Munuera J, Domenech S, Erickson KI, Mataro M. Effects and Mechanisms of Cognitive, Aerobic Exercise, and Combined Training on Cognition, Health, and Brain Outcomes in Physically Inactive Older Adults: The Projecte Moviment Protocol. Front Aging Neurosci. 2019 Aug 14;11:216. doi: 10.3389/fnagi.2019.00216. eCollection 2019. PMID 31481889
- See also: blog of the project — http://projectemovimentblog.wordpress.com/portfolio/priojecte-1/
- See also: Neuroscience Institute University of Barcelona — http://www.neurociencies.ub.edu/en/
- See also: IDIAP Jordi Gol — http://www.idiapjordigol.com/